CLINICAL TRIAL: NCT06470984
Title: Ethics Education Supporting Acute and Post-Acute Nurse Leaders - 2nd Cohort
Brief Title: Ethics Education to Support Nurse Leaders in HealthCare
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Jill K. Greenwood-Williamson, Director of Clinical Education, OSF Healthcare System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2193504
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: nursing ethics; clinical ethics; ethical competence
MeSH Terms: conditions — Behavior | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acute Care (Experimental): Nursing leaders will participate voluntarily and will report their leadership role as acute care (hospital settings).
  Interventions: Behavioral: Educational intervention
- Post-Acute Care (Experimental): Nursing leaders will participate voluntarily and will report their leadership role as post-acute care (ambulatory settings)
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — Professional development program provided online to small groups of professional nurse leaders via an educational platform over a 6-week period.

SUMMARY:
Using an exploratory study design with an educational intervention, a pre/post evaluation of ethical confidence and competence will be completed for nursing leaders working in either acute care or post-acute care with primary purpose to increase ethical competency and confidence in decision making for nursing leaders in a clinical role.

DETAILED DESCRIPTION:
The purpose of this project is to implement an ethics educational program that has been developed in collaboration with subject matter experts to support patient facing nursing leaders. The intervention is an ethics education pathway, which will be used for approximately 60-80 patient-facing nurse leaders who practice in either acute care or post-acute care over a 6-week period. One Pre and two post-assessment questionnaires will be distributed, which include the "Ethical Competence Support Questionnaire" © and the "Ethical Safety Questionnaire" ©. Permission for the instrument use was obtained from the author.

ELIGIBILITY:
Inclusion Criteria:

* employment within an in-patient or outpatient non-profit healthcare setting as a nursing leader.
* settings include acute-care units and post-acute care facilities

Exclusion Criteria:

* nurses working direct care 100% of their time without any formal leadership responsibilities

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ethical Competence Support Questionnaire | change from baseline in the ethical competence measure at 6 weeks after initiation.
  The ethical competence support questionnaire contains 27 items addressing four subcategories: encouragement of ethical activity, provision of information on ethical issues, dealing with ethical issues, and conversational support. A 5-point Likert Scale is used for measurement: Strong disagree to Strongly Agree. Minimum value = 1 maximum value =5.
Ethical Safety Questionnaire | change from baseline in the ethical safety measure at 6 weeks after initiation.
  The ethical safety questionnaire contains11 items addressing four subcategories: general ethical safety, ethical autonomy, ethical respect, and ethical competence. A 5-point Likert Scale is used for measurement: Strong disagree to Strongly Agree. Minimum value = 1 maximum value =5.

SECONDARY OUTCOMES:
Ethical Confidence Assessment | change from baseline in the ethical competence measure at 6 weeks following initiation and at 3 months.
  Confidence as a nurse leader for ethical decision making is rated on a 1-10 scale. 0=not confident 10= very confident

CONTACTS AND LOCATIONS:
Overall Officials: Jill K Greenwood-Williamson, DNP, RN, Principal Investigator — OSF HealthCare
Locations (1):
- OSF HealthCare, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aitamaa E, Suhonen R, Iltanen S, Puukka P, Leino-Kilpi H. Ethical problems in nursing management: Frequency and difficulty of the problems. Health Care Manage Rev. 2021 Jan/Mar;46(1):25-34. doi: 10.1097/HMR.0000000000000236. PMID 30724758
- [Background] Barkhordari-Sharifabad M, Ashktorab T, Atashzadeh-Shoorideh F. Obstacles and problems of ethical leadership from the perspective of nursing leaders: a qualitative content analysis. J Med Ethics Hist Med. 2017 Feb 21;10:1. eCollection 2017. PMID 28523116
- [Background] Poikkeus T, Suhonen R, Katajisto J, Leino-Kilpi H. Organisational and individual support for nurses' ethical competence: A cross-sectional survey. Nurs Ethics. 2018 May;25(3):376-392. doi: 10.1177/0969733016642627. Epub 2016 May 10. PMID 27165144
- [Background] Poikkeus T, Suhonen R, Katajisto J, Leino-Kilpi H. Relationships between organizational and individual support, nurses' ethical competence, ethical safety, and work satisfaction. Health Care Manage Rev. 2020 Jan/Mar;45(1):83-93. doi: 10.1097/HMR.0000000000000195. PMID 29533273
- [Background] Salmela S, Koskinen C, Eriksson K. Nurse leaders as managers of ethically sustainable caring cultures. J Adv Nurs. 2017 Apr;73(4):871-882. doi: 10.1111/jan.13184. Epub 2016 Nov 11. PMID 27732746